CLINICAL TRIAL: NCT06467747
Title: The Efficacy of Intraoperative Music Stimulation on Perioperative Pain Management
Brief Title: The Efficacy of Music on Perioperative Pain Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Tzu Chi Hospital (Other)
Responsible Party: Principal Investigator, Sih-hua Chen, Attending Physician, Department of Anesthesiology, Taichung Tzu Chi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC113-11
Record Dates: First submitted 2024-06-12; First posted 2024-06-21 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Perioperative Pain Management
Keywords: Music therapy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music group (Experimental): Listen music with earphone
  Interventions: Other: Music
- Mute group (Placebo Comparator): Keep mute under earphone
  Interventions: Other: Mute
- Control group (No Intervention): As usual anesthesia care without earphones

INTERVENTIONS:
Other: Music — Music group: wear earphones to listen to music and receive standardized anesthesia protocol
  Arms: Music group
Other: Mute — Mute group: wear earphones without music and receive standardized anesthesia protocol
  Arms: Mute group

SUMMARY:
The goal of this clinical trial is to learn if intraoperative music stimulation works to alleviate perioperative pain in surgical patients undergoing general anesthesia. It will also learn about the possible mechanisms by how music affects pain.

The main questions it aims to answer are:

Does music lower the number of times participants need to use a rescue analgesic? What changes occur in electroencephalogram (EEG) and nociception monitors when participants listen to music? Researchers will compare music to mute or control (hear ambient sounds without earphones) to see if music works to alleviate perioperative pain.

Participants will listen music or mute or ambient sounds throughout the operation, and receive routine anesthesia care.

ELIGIBILITY:
Inclusion Criteria:

* Older than 20 years old and younger than 80 years old
* male or female
* Scheduled for minimally invasive surgery (laparoscopic cholecystectomy, appendectomy)
* Ambulatory surgery
* American Society of Anesthesiologists (ASA) physical status I~III

Exclusion Criteria:

* Severe hearing impairment
* Severe pulmonary or cardiovascular disease
* Brain or central nervous system (CNS) disorder
* Long-term systemic steroid or daily morphine treatment
* Pregnant women
* Emergency surgery
* The absence of informed consent

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | 1. While in the post-anesthesia care unit, for an average of 1 hour. 2. 24 hours after surgery.
  To assess pain severity using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable". Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
Analgesic-frequency | 1. During the operation. 2. While in the post-anesthesia care unit, for an average of 1 hour. 3. 24 hours after surgery.
  Frequency of analgesic usage
Analgesic-total amount | 1. During the operation. 2. While in the post-anesthesia care unit, for an average of 1 hour. 3. 24 hours after surgery.
  Total amount of analgesic used
Post-operative nausea and vomiting (PONV) | 1. While in the post-anesthesia care unit, for an average of 1 hour.
  Frequency of nausea and vomiting episodes

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Ling Shen, Principal Investigator — Taichung Tzu Chi Hospital
Locations (1):
- Taichung Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Taichung, Not in USA, Taiwan

IPD SHARING:
Plan to Share IPD: No